CLINICAL TRIAL: NCT05666895
Title: Role of CBC as a Prognostic Marker for DKA Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Tawfik Abdelaleem, Resident, Assiut University
Other Study IDs: CBC in DKA Patients
Record Dates: First submitted 2022-12-14; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Diabetic Ketoacidosis
Keywords: CBC in DKA Patients
MeSH Terms: conditions — Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To evaluate that change of platelet-to-lymphocyte Ratio affect the duration of hospital stay and mortality rate of DKA patients
2. To assess the impact of red blood cell distribution width (RDW) on the prognosis of diabetic ketoacidosis patients
3. To evaluate the changes in hematological parameters (RBCs,Hct,Hb,MCV,PLT,WBCs) and their correlations with acidosis level and dehydration during ketoacidosis treatment

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a serious threat to global health with an increasing prevalence and incidence rates,The number of people who had DM was 463 million in 2019,and according to international diabetes federation [IDF] this number will have reached 700 million in 2045 (1).

One of the most serious complication of DM is diabetic ketoacidosis (DKA) which is a life-threatening acute copmlication of diabetes mellitus [DM], [DKA] occur in patients with both type 1 and type 2 diabetes, for which type 1 and type 2 diabetes is responsible for 66% and 34% patients respectively (2,3).

Despite the development of improved treatment, DKA remains at a high incidence of recurrence and a leading cause of mortality among patients with DM, resulting in an elevated burden for patients,hospitals,and healthcare providers(4,5).

As a systemic metabolic disease,DKA has been reported to be associated with the inflammatory response of the hyperglycaemic state(6,7). the inflammatory markers like (platelets-lymphocyte ratio, red blood cell distribution width) play an important role in the development of inflammation and affect prognosis of DKA One of the most things that affected by diabetic ketoacidosis is hydration status, As DKA can cause dehydration and some complications may result from that such as cerebral edema,coma or even death(8,9).

there are many methods to estimate the hydration status such as clinical dehydration scale(CDS), hematological parameters (RBC, Hct , Hb MCV, PLT ,WBC) which are used as an alternative approach to estimate the extent of dehydration in DKA patients(10,11).

ELIGIBILITY:
Inclusion Criteria:

* The study will include patient with type 1 or type 2 DM, patients > 18 yrs, DKA patients (based on the criteria of the American Diabetes Association (ADA): plasma glucose > 13.9 mmol/l (250 mg/dL), arterial pH < 7.3 and a bicarbonate level <18 mEq/l, with ketonuria)

Exclusion Criteria:

* The study will exclude patients <18 yrs , patients with history of hematological disease like(leukemia,hemophilia,thalassemia,sickle cell anaemia,polycythemia vera),patients with history of renal or cardiac or hepatic disease)

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Patients admitted at ICU at internal medicine departement from 1/2023 to 6/2024
  2. Complete history and through clinical examination and investigations at admission and discharge
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Measure of inflammatory markers like (platelets-lymphocyte ratio, red blood cell distribution width) changes in DKA patients and affection of these changes on inflammation development and prognosis of DKA | Baseline
  the inflammatory markers like (platelets-lymphocyte ratio, red blood cell distribution width) play an important role in the development of inflammation and affect prognosis of DKA and and changes in these markers also affect duration of hospital stay and mortality rate in DKA patients

SECONDARY OUTCOMES:
Hematological parameters (RBC, Hct , Hb MCV, PLT ,WBC) which are used as an alternative approach to estimate the extent of dehydration in DKA patients | Baseline
  there are many methods to estimate the hydration status such as clinical dehydration scale(CDS), hematological parameters (RBC, Hct , Hb MCV, PLT ,WBC) which are used as an alternative approach to estimate the extent of dehydration in DKA patients

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine assuit university, Asyut, Egypt

REFERENCES:
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2014 Jan;37 Suppl 1:S81-90. doi: 10.2337/dc14-S081. No abstract available. PMID 24357215
- [Background] Seth P, Kaur H, Kaur M. Clinical Profile of Diabetic Ketoacidosis: A Prospective Study in a Tertiary Care Hospital. J Clin Diagn Res. 2015 Jun;9(6):OC01-4. doi: 10.7860/JCDR/2015/8586.5995. Epub 2015 Jun 1. PMID 26266145
- [Background] Misra S, Oliver N, Dornhorst A. Diabetic ketoacidosis: not always due to type 1 diabetes. BMJ. 2013 Jun 10;346:f3501. doi: 10.1136/bmj.f3501. No abstract available. PMID 23751904
- [Background] Lohiya S, Kreisberg R, Lohiya V. Recurrent diabetic ketoacidosis in two community teaching hospitals. Endocr Pract. 2013 Sep-Oct;19(5):829-33. doi: 10.4158/EP13057.RA. PMID 23757621
- [Background] Zargar AH, Wani AI, Masoodi SR, Bashir MI, Laway BA, Gupta VK, Wani FA. Causes of mortality in diabetes mellitus: data from a tertiary teaching hospital in India. Postgrad Med J. 2009 May;85(1003):227-32. doi: 10.1136/pgmj.2008.067975. PMID 19520872
- [Background] Xu L, Wang L, Huang X, Liu L, Ke W, He X, Huang Z, Liu J, Wan X, Cao X, Li Y. Baseline red blood cell distribution width predicts long-term glycemic remission in patients with type 2 diabetes. Diabetes Res Clin Pract. 2017 Sep;131:33-41. doi: 10.1016/j.diabres.2017.06.019. Epub 2017 Jun 15. PMID 28672172
- [Background] Li W, Huang E, Gao S. Type 1 Diabetes Mellitus and Cognitive Impairments: A Systematic Review. J Alzheimers Dis. 2017;57(1):29-36. doi: 10.3233/JAD-161250. PMID 28222533
- [Background] Wolfsdorf JI, Glaser N, Agus M, Fritsch M, Hanas R, Rewers A, Sperling MA, Codner E. ISPAD Clinical Practice Consensus Guidelines 2018: Diabetic ketoacidosis and the hyperglycemic hyperosmolar state. Pediatr Diabetes. 2018 Oct;19 Suppl 27:155-177. doi: 10.1111/pedi.12701. No abstract available. PMID 29900641
- [Background] Bruck E. Laboratory tests in the analysis of states of dehydration. Pediatr Clin North Am. 1971 Feb;18(1):265-83. doi: 10.1016/s0031-3955(16)32538-x. PMID 25868190
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249